CLINICAL TRIAL: NCT06014346
Title: Prospective Study of the Prevention of Vasovagal Reactions in First-time Whole Blood Donors Using a Combined PSYchological and Physiological Approach: PREDONPSY
Brief Title: Prevention of Vasovagal Reactions in First-time Blood Donors Using a Combined PSYchological and Physiological Approach
Acronym: PREDONPSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL22_0131
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Vasovagal Reaction
Keywords: first time donor; whole blood donation; vasovagal Reaction; physiological; psychological; BDRI; BDAS
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): EFS usual standard practices for the whole blood donation
- Test Group 1 (Experimental): A psychological strategy is added to EFS standard practices before the whole blood donation
  * flyer given at the interview presenting the 4 most frequent fears as well as a description of the recommended muscular and breathing exercises,
  * followed by a training of these exercises and their execution
  Interventions: Other: Psychological strategy
- Test Group 2 (Experimental): A physiological strategy is added to EFS standard practices before the whole blood donation : - Ingesting a salty snack.
  Interventions: Other: Physiological strategy
- Test group 3 (Experimental): The both psychological and physiological strategies are added to EFS standard practices before the whole blood donation
  * flyer given at the interview presenting the 4 most frequent fears as well as a description of the recommended muscular and breathing exercises,
  * followed by a training of these exercises and their execution Ingesting a salty snack.
  Interventions: Other: Psychological strategy; Other: Physiological strategy

INTERVENTIONS:
Other: Psychological strategy — * flyer given at the interview presenting the 4 most frequent fears as well as a description of the recommended muscular and breathing exercises,
  * then realization accompanied by a training of these exercises
  Arms: Test Group 1; Test group 3
Other: Physiological strategy — - ingesting a salty snack
  Arms: Test Group 2; Test group 3

SUMMARY:
The prevention of vasovagal reactions (VVR) occurring during or after donation is a major issue for the French Blood Establishment (EFS), firstly to guarantee the safety of donors but also to retain them, as this reaction is one of the negative experiences affecting the return to donation.

The EVASION study conducted in the Auvergne Rhône-Alpes region (AURA) on 4828 donors representative of the French donor population, reported a beneficial effect of muscle contraction exercises to prevent the occurrence of VVR during donation, while hydric solutions, and even more so isotonic solutions, were likely to decrease the frequency of delayed VVR.

These preventive measures have been integrated into the internal guidelines and currently include muscular and breathing exercises and hydration. Nevertheless, the isotonic solution could not be routinely deployed for feasibility and cost reasons. A salty snack could replace the isotonic solution to produce the same effects with better feasibility and acceptability. Furthermore, a significant proportion of discomfort is psychological in origin, related to stress and anxiety which persist despite these measures, particularly in the first-time donor population.

These measures, which are mainly focused on the prevention of VVR of physiological origin, are still insufficient and can be optimized and complemented to reduce the occurrence of VVR, especially in first-time donors for whom anxiety and stress play an important role in the etiology of VVR.

Two measures could further reduce the occurrence of VVR:

* Reinforcement of the physiological strategy: ingestion of a salty snack before donation, the effect of which could be similar to the effect of the isotonic solution, which could not be delivered in practice because of its cost following the data of the EVASION study.
* Addition of a psychological strategy: flyer given at the interview presenting the four most frequent fears as well as a description of the recommended muscular and respiratory exercises, followed by the execution of the recommended exercises before the sampling.

Hypothesis is that the combination of a psychological and physiological strategies would allow a reduction of the occurrence of immediate and/or 48 h delayed VVR during the whole blood donation in first time donors compared to the current practices.

ELIGIBILITY:
Inclusion Criteria:

* M/F between 18 and 70 years old,
* A first-time donor who wishes to donate blood in Lyon, either at a fixed site or at a mobile unit,
* Declared fit to donate whole blood after the EFS pre-donation interview,
* Weight ≥ 50kg and height ≥ 135 cm,
* Available for telephone contact between to 5d +/- 2 days after donation,
* Having signed a written consent to participate in the study.

Non-inclusion criteria:

* Known allergy to shellfish, and/or gluten, and/or milk, and/or soy,
* Incomprehension of the French language,
* First-time donor under protective measures (guardian, curator) or any other administrative measure,
* Not affiliated to the French social security system or any other equivalent system,
* Pregnant or breastfeeding woman,
* Subject participating in any other interventional or non-interventional research

Exclusion Criteria:

* Withdrawal of consent
* First-time donor with anemia following routine hemoglobin testing
* First-time donor not reachable for telephone interview

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5320 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2025-05-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Vasovagal reactions (VVR) | Day 1 = donation day ; Day 3 = 48h post donation
  Proportion of first-time donors experiencing VVR (immediate and delayed up to 48 hours) during whole blood donation managed by both psychological and physiological strategies (group 4) compared to usual standard practices (group 1)

SECONDARY OUTCOMES:
VVR psychological strategy | Day 1 = donation day ; Day 3= 48h post donation
  Proportion of first-time donors experiencing VVR (immediate and delayed up to 48 hours) during whole blood donation managed by psychological strategy (group 2) compared to usual standard practices (group 1)
VVR physiological strategy | Day 1 = donation day ; Day 3= 48h post donation
  Proportion of first-time donors experiencing VVR (immediate and delayed up to 48 hours) during whole blood donation managed by physiological strategy (group 3) compared to usual standard practices (group 1)
Immediate VVR | Day 1 = donation day, before leaving the centre
  Proportion of first-time donors with immediate VVR compared between the groups
Delayed VVR | Day 3= 48h post donation
  Proportion of first-time donors with delayed VVR compared between the groups
First-time donor adherence | Day 1 = donation day, before leaving the centre
  Adherence of the primary donor to the study strategies and to the EFS recommendations (complete intake of salty snacks, hydration, performance of muscle and breathing exercises training, performance of muscle and breathing exercises during donation, compliance with the duration of post-donation monitoring stage).
Anxiety/fear | Day 1 = donation day, before donation
  Assessment of the evolution of the "anxiety/fear" score between arrival and before the whole blood donation, compared between the groups.
  This questionnaire consists of the 6-item Blood Donor Anxiety Scale (BDAS) (5-point Likert scale) (Chell et al., 2016) and a 4-item component with a 5-point Likert scale that allows for an assessment of the 4 most common donor fears (of the needle, to see blood, to feel pain, to experience sensations of discomfort). The scoring is obtained by summing up the responses to the different items.
  Score is between 10 and 50, a higher score is associated to a better outcome.
Sense of control and fears | Day 1 = donation day, before donation
  Assessment of the "sense of control and fears" score, compared between the groups.
  The concepts measured here are the feeling of control related to giving blood (5 items) and the feeling of control over fears (4 items) according to a 5-point Likert scale. The scoring is obtained by summing up the answers to the different items.
  Score is between 9 and 45, a higher score is associated to a better outcome.
Feelings of discomfort | Day 1 = donation day, after donation and before leaving the centre
  Assessment of the "feelings of discomfort" score, compared between the groups. The BDRI (Blood Donation Reactions Inventory) (France et al., 2008) provides an assessment of the subjective evaluation of 11 pre-syncopal symptoms (5-point Likert scale). The BDRI is easily understood by donors and is rapid. The BDRI provides important information about the donor experience to predict satisfaction and likelihood of re-donation. The score is calculated by summing up the responses to the various items.
  Score is between 11 and 55, a higher score is associated to a worse outcome.
First-time donor retention | Month 12 following the first-time donation
  Compared between the groups the number of first-time donors who made a second blood donation in the 12 months following the first-time donation, collected by query from the EFS computerized file

CONTACTS AND LOCATIONS:
Locations (1):
- French Blood Establishment (EFS), Lyon, France

IPD SHARING:
Plan to Share IPD: No